CLINICAL TRIAL: NCT01924052
Title: CGRP Induced Migraine Attacks in Patients With High and Low Genetic Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, MD, Danish Headache Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-2-2011-141
Record Dates: First submitted 2013-08-10; First posted 2013-08-16 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Calcitonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Migraine patients with high genetic load (Active Comparator): CGRP intravenous infusion 1.5 microgram/min for 20 min
  Interventions: Drug: CGRP
- Migraine patients with low genetic load (Active Comparator): CGRP intravenous infusion 1.5 microgram/min for 20 min
  Interventions: Drug: CGRP

INTERVENTIONS:
Drug: CGRP — Calcitonin-gene-related-peptide (CGRP)
  Other Names: calcitonin-gene-related peptide

SUMMARY:
The investigators hypothesized that migraine without patients with many genetic loci associated with migraine (high genetic load) would be more sensitive and get provoked more migraine attacks by calcitonin gene-related peptide (CGRP) compared to patients with few genetic loci associated with migraine (low genetic load).

DETAILED DESCRIPTION:
Migraine is a very prevalent neurological disorder with a strong genetic factor. The common forms of migraine have a multifactorial and polygenic pattern of inheritance and genetics research is crucial for a deeper understanding of migraine mechanisms. Recently, 12 genetic loci have been identified to be associated with migraine with (MA) and without aura (MA) in four large genome-wide association studies (GWAS). The functional consequences of these genetic loci in humans are yet unknown.

Calcitonin gene-related peptide (CGRP) is a neuropeptide which plays a crucial role in the pathophysiology of migraine and is present in migraine relevant structures. CGRP can induce migraine attacks in MO patients via an adenosine monophosphate (cAMP) dependent pathway and CGRP antagonism is efficient in the treatment of migraine attacks. Also, a recent study has showed that intracellular accumulation of cAMP is crucial for the induction of migraine attacks. However, CGRP does not cause migraine attacks in familial hemiplegic migraine (FHM), an autosomal dominant subtype of MA.

The phenotype of the migraine inducing effects of CGRP might therefore be linked to some of the 12 genetic susceptibility loci that have been identified. One of the genetic loci (rs13208321) is located in a gene (FHL5) that is associated with the regulation of cAMP-responsive elements.

ELIGIBILITY:
Inclusion Criteria:

- Migraine without aura patients genotyped for the 12 newly idetified gene variants associated with migraine.

Exclusion Criteria:

* Other primary headache
* A history of cerebrovascular disease and other CNS- disease
* A history suggesting ischaemic heart disease
* Serious somatic and mental disease
* Hypo- or hypertension
* Abuse of alcohol or medicine (opioid analgesics).
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
CGRP induced migraine attacks in patients with high and low genetic load | Change from baseline in headache intensity at 12 hours after the start of infusion of CGRP
  The difference in incidence of migraine-like attacks between patients with high genetic load and patients with low genetic load using verbal rating scale (VRS).

SECONDARY OUTCOMES:
CGRP induced migraine attacks in patients with high and low genetic load | Change from baseline in headache intensity at 12 hours after the start of infusion of CGRP
  The difference in area under the curve (AUC) for headache intensity scores (0-12 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Song Guo, MD, Principal Investigator — Danish Headache Center & Department of Neurology